CLINICAL TRIAL: NCT01397292
Title: Registry Examining Retrospective and Prospective Data for Patients Undergoing Pulmonary Procedures
Brief Title: Registry for Patients Undergoing Pulmonary Procedures
Status: Terminated | Type: Observational
Why Stopped: funding/ enrollment
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM13603
Record Dates: First submitted 2011-07-15; First posted 2011-07-19 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2011-07

CONDITIONS: Pulmonary Procedures
Keywords: Bronchoscopy; Interventional Pulmonary; Pleuroscopy; Tracheostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to examine the safety, tolerability, and effectiveness of currently available pulmonary procedures when used to diagnose or treat different diseases.

This study will collect information that may influence the outcome of the procedure and identify factors that may affect the procedures yield or safety. The information will be entered into a registry or data storage.

DETAILED DESCRIPTION:
This is a retrospective and prospective data registry of all pulmonary diagnostic and therapeutic interventional pulmonary procedures at a single academic center. All pulmonary procedures upon completion will be entered into a database by the participating investigator performing the procedure. For both diagnostic and therapeutic cases, the data will require additional input 1-4 weeks after the procedure in order to place the diagnosis and follow-up data. Retrospective data will only be collected for patients that had their procedures prior to approval of this registry.

Study data will be collected and managed using REDCap (Research Electronic Data Capture) electronic data (CTSA Awared - Award Number UL1RR031990) capture tools hosted at Virginia Commonwealth University. REDCap is a secure, web-based application designed to support data capture for research studies.

The prison population will also be included in the registry in order to examine the effects of pulmonary procedures on a special population.

ELIGIBILITY:
Inclusion Criteria:

* ADULT PATIENTS (>18 YEARS OLD) that have a planned PULMONARY PROCEDURE

Exclusion Criteria:

* ALL KNOWN PREGNANT PATIENTS WILL BE EXCLUDED FROM THIS REGISTRY.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ONLY ADULT PATIENTS (>18 YEARS OLD) that have a planned PULMONARY PROCEDURE will be potential participants. This will also include a special group, prisoners.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2011-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans J Lee, M.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States